CLINICAL TRIAL: NCT01024634
Title: Vascular and Neuro-inflammatory Effects of Endurance Exercise Training in African Americans
Acronym: VINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bo Fernhall, Professor, University of Illinois at Urbana-Champaign
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UIUC 09599; 1R01HL093249-01A1 (NIH)
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Vascular Health; Autonomic Function
Keywords: Arterial stiffness; Endothelial function; Autonomic function; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- African American Group (Other): A group of young African American males and females
  Interventions: Behavioral: Endurance Exercise
- Caucasian Group (Other): a group of young Caucasian men and women
  Interventions: Behavioral: Endurance Exercise

INTERVENTIONS:
Behavioral: Endurance Exercise — 8 weeks of Endurance exercise training, 3-4 times per week, 45-60 minutes perr session

SUMMARY:
The purpose of this study is to test the effects of endurance exercise training on arterial structure and function, and to examine potential mechanisms producing changes in arterial structure and function in young (18-35 years of age) African Americans when compared to Caucasians.

DETAILED DESCRIPTION:
African-Americans are at greater risk than Caucasians for developing hypertension, cardiovascular disease, stroke and renal disease. This is likely related to arterial dysfunction including greater arterial stiffness, and reduced microvascular reactivity of resistance arteries in African-Americans. In addition, African-Americans have higher levels of inflammatory markers, and a greater sympathoexcitatory response to various stressors. This imbalance between sympathetic and reduced parasympathetic activation may directly affect vascular function and potentiate a greater inflammatory response, further altering key structural and functional properties of the vascular wall. The overall aim of this proposal is to test the effects of endurance exercise training on arterial structure and function, and to examine potential mechanisms producing changes in arterial structure and function in young (18-35 years of age) African Americans when compared to Caucasians. We will examine these effects at rest and following a high intensity (maximal cycle ergometry) sympathoexcitation at both pre- and post-intervention time points, since sympathoexcitation may elucidate changes not evident at rest. Because African-Americans have higher levels of arterial stiffness, lower microvascular reactivity, greater responses to sympathoexcitation, greater levels of inflammatory markers and greater vasoconstrictive tone, we hypothesize that African-Americans will show differential responses to exercise training and benefit more compared to a matched group of Caucasians.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in good health with no cardiovascular, metabolic, or inflammatory disease, who do not use cardiovascular medications or antioxidant vitamin supplementation, including use of anti-inflammatory (including aspirin) or steroidal substances in the past 2 months will be inlcuded

Exclusion Criteria:

* Subjects who smoke, are severely obese (body mass index > 35 kg/m2), or who have hypertension (blood pressure >140/90mmHg), diabetes (fasting glucose >110mg/dl), hyperlipidemia, inflammatory disease (rheumatoid arthritis and systemic lupus erythematosus, etc) or diagnosed cardiovascular disease including, coronary heart disease, hypertension and cardiac arrhythmia or renal disease, will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Arterial function | Pre, following a 4 week control period and after 8 weeks of exercise intervention

SECONDARY OUTCOMES:
Autonomic function | Pre, following a 4 week control period and following 8 weeeks of an exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fernhall, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Kinesiology and Community Health Department, University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Derived] Maroco JL, Lane AD, Ranadive SM, Yan H, Baynard T, Fernhall B. Aerobic Training Attenuates Differences Between Black and White Adults in Left Ventricular-Vascular Coupling and Wasted Pressure Effort. J Am Heart Assoc. 2024 Nov 5;13(21):e036107. doi: 10.1161/JAHA.124.036107. Epub 2024 Nov 4. PMID 39494565